CLINICAL TRIAL: NCT02319109
Title: A Prospective, Single-Center Study, in Healthy Volunteers to Establish a PT/INR Reference Interval for the Microvisk INR Test System
Brief Title: PT/INR Reference Interval IN Healthy Volunteers
Acronym: REF01
Status: Completed | Type: Observational
Sponsor: Microvisk Technologies Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: 2011/REF01
Record Dates: First submitted 2014-12-09; First posted 2014-12-18 (Estimated); Last update posted 2015-01-22 (Estimated); Status verified 2014-12

CONDITIONS: Healthy

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a prospective, single-center study in healthy volunteers to establish a PT/INR reference interval for the Microvisk International Normalized Ratio (INR) Test System. The primary objective of this study is to establish the reference interval for the measurement of prothrombin time (PT/INR) using the Microvisk INR Test System. The second objective is to evaluate the safety of the device.

DETAILED DESCRIPTION:
Healthy volunteers who meet eligibility criteria, have been fully informed and provided written informed consent will be enrolled into this study. Each participant will be required to donate up to 3 finger stick samples for testing on one occasion. The maximum trial duration for each participant is one visit/occasion. This will be followed by a standard venipuncture for (1) a neutral tube (Red Top) for analysis by the on-test method, (1) one sodium citrate tube (Blue Top) for analysis by the comparative/reference laboratory method. Sample collection will take place within the clinic session. The maximum trial duration for each participant is one clinic session.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is considered a healthy volunteer
2. Subject is male or female, over 18 years of age
3. Subject is informed and has been given ample time and opportunity to think about his/her participation and has given his/her written informed consent
4. Subject agrees to have blood drawn (venipuncture) and finger stick

Exclusion Criteria:

1. Subject is unable to give informed consent
2. Subject is less than 18 years of age
3. Female subject is pregnant
4. Subject is on anticoagulant medication or other medication known to affect PT/INR assessment (e.g., warfarin, heparin) for a minimum of 28 days before enrolling in the trial
5. Subject has a medical condition known to affect PT/INR (e.g. vitamin K deficiency, disseminated intravascular coagulation, liver disease, decreased or defective factor I, II, V, VII, or X)
6. Subject has already taken part in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy male and female subjects, not taking any oral vitamin K antagonist therapy, over the age of 18 years.
Sampling Method: Non-Probability Sample
Enrollment: 154 (Actual)
Dates: Start 2014-12; Primary Completion 2014-12 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
INR value for normal population | 1 day
  Establish the INR value for the normal population

SECONDARY OUTCOMES:
Safety (Number of Participants with Adverse Events) | 1 day
  Number of Participants with Adverse Events as a Measure of Safety
Device Failure (number of device failures) | up to 12 weeks
  Overall number of device failures to measure the robustness of system

CONTACTS AND LOCATIONS:
Overall Officials: Helen Stacey, MD, PhD, Principal Investigator — Diablo Clinical Research
Locations (1):
- Diablo Research Clinic, Walnut Creek, California, United States